CLINICAL TRIAL: NCT00419432
Title: Functional Outcomes Following Orthopaedic Surgery Based on Gait Laboratory Versus Observational Gait Analysis in Ambulatory Children With Cerebral Palsy: A Multi-center Randomized Controlled Trial.
Brief Title: Outcomes of Orthopaedic Surgery Using Gait Laboratory Versus Observational Gait Analysis in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Unni Narayanan, Orthopaedic Surgeon, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000009387
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
Keywords: Pediatrics; Cerebral Palsy; Gait Analysis; Orthopedic Surgery
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (standard pre-operative analysis) (Active Comparator)
  Interventions: Other: Routine Observational Analysis (prior to procedure)
- Group B (additional pre-operative analysis) (Experimental)
  Interventions: Other: Routine Observational analysis supplemented with Gait Lab Information (prior to procedure)

INTERVENTIONS:
Other: Routine Observational Analysis (prior to procedure) — Controls will undergo the standard orthopaedic surgery using the information from the physical examination and observational analysis of the gait alone.
  Arms: Group A (standard pre-operative analysis)
Other: Routine Observational analysis supplemented with Gait Lab Information (prior to procedure) — This experimental group will undergo standard orthopaedic surgery using the information from the physical examination, observational AND the gait laboratory analysis data
  Arms: Group B (additional pre-operative analysis)

SUMMARY:
The purpose of this pilot trial is to determine whether the addition of gait laboratory analysis for surgical decision making, compared with the use of observational analysis alone, results in improved functional outcomes in ambulatory children with cerebral palsy undergoing multi-level lower extremity orthopaedic surgery.

DETAILED DESCRIPTION:
Children with cerebral palsy, who are ambulatory, have an inefficient gait often associated with functional disability. Many of these children are candidates for orthopaedic surgery, which includes multi-level soft tissue and bony procedures. Pre-operative planning is based on the physical examination and visual (observational) analysis of the child's gait. In some centres, patients undergo additional gait analysis in a motion laboratory. While gait laboratory analysis is accepted as an important research tool, there is controversy about its clinical utility in decision making for the surgical management of this population. To date, no clinical trials have been undertaken to answer this question, and the appropriate clinical utilization of this technology is yet to be established. The consequence of this uncertainty is that ambulatory children with cerebral palsy are either being deprived of a useful assessment tool in some centres, or alternatively they are being subjected to an unnecessary evaluation that is both expensive and time consuming in other centres. A multi-centre randomized trial will provide evidence to support or refute the need for gait laboratory analysis for surgical decision-making for this population. This pilot randomized controlled trial in four sites will assess the feasibility of, and provide the template for the design and conduct of the definitive larger multi-centred trial to extend its generalizability across North America and other jurisdictions. The specific objectives include:

1. Establish the feasibility of implementing the randomized trial study design in multiple centres
2. Estimate recruitment rates and timelines
3. Establish responsiveness of outcome measures to finalize the primary & secondary outcomes
4. Estimate effect sizes of functional outcomes for sample size calculations
5. Establish data management system (web-based database) for definitive multi-centre study.
6. Assess feasibility, reliability and face validity of pilot health economic data forms to include health economic evaluation in the future definitive multi-centre trial.

   Secondary objectives include:
7. Does the addition of gait analysis alter surgical decisions made from video observation alone, when performed in the setting of this pilot trial?
8. Evaluate the consistency of the surgical decision making: intra- & inter rater reliability

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of spastic cerebral palsy.
2. Age 6 to 15 years at the time of the initial assessment.
3. Gross Motor Function Classification System (GMFCS) levels II or III (demonstrable independent ambulatory potential with or without orthotics/assist devices).
4. Patients have been referred for assessment and treatment of gait abnormality.
5. Patients have a gait abnormality interfering with their physical function.
6. Patients are candidates for orthopaedic surgery including soft tissue and/or bony procedures involving at least 2 levels, in one or both lower extremities (e.g. knee & ankle).
7. Patients must be able to undergo instrumented gait analysis in a motion laboratory.

Exclusion Criteria:

1. Presence of dystonia, athetosis, or mixed tone abnormalities.
2. History of orthopaedic lower extremity procedures within the previous 2 years.
3. Patients who have had previous gait laboratory analysis that has been seen by the treating surgeon.
4. Patients who will be unable to return for the required follow up visits/gait analysis.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2019-08 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
General Effect Size of Secondary Outcomes | Post Study
  The final primary and secondary outcome measures will be chosen based on responsiveness and their effect sizes used to calculate sample size for a future definitive trial.

SECONDARY OUTCOMES:
Gross Motor Function Measure (GMFM-66) | Baseline, 6, 12, 24 months follow up
  A well validated condition specific clinical measure to evaluate change in motor function in children with cerebral palsy
Pediatric Outcomes Data Collection Instrument(PODCI) | Baseline, 6, 12, 24 months follow up
  A generic measure of musculoskeletal functional health outcomes in children and adolescents
Gillette Functional Assessment Questionnaire (FAQ) | Baseline, 6, 12, 24 months follow up
  A validated condition specific functional walking scale developed for children with cerebral palsy
Functional Mobility Scale (FMS) | Baseline, 6, 12, 24 months follow up
  Developed to measure functional mobility of a child in three different environments (home, school, and the wider community).
Activity Scale for Kids (ASK) | Baseline, 6, 12, 24 months follow up
  A reliable and valid, self-report measure of childhood physical disability.
Gillette Gait (Normalcy) Index (GGI) | Baseline, 6, 12, 24 months follow up
  Quantifies the magnitude of gait deviation from normal
Gait Parameters | Baseline, 12-, 24-months follow-up
  Gait velocity; Stride length; O2 consumption & O2 Cost during walking

CONTACTS AND LOCATIONS:
Overall Officials: Unni Narayanan, MBBS, MSc, FRCSC, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (6):
- Canada (6):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - British Columbia's Children's Hospital, Vancouver, British Columbia
  - Erinoak Centre, Mississauga, Ontario
  - Grandview Children's Rehabilitation Centre, Oshawa, Ontario
  - Bloorview Kids Rehab, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario